CLINICAL TRIAL: NCT00064402
Title: A Double-Blind, Double-Dummy, Randomized, Placebo- and Active-Controlled, Multicenter, Parallel-Group Study of (R,R)-Formoterol in the Treatment of Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: Determine the Safety and Efficacy of (R,R)-Formoterol in the Treatment of Subjects With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 091-051
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Chronic Bronchitis; Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — Formoterol Fumarate; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): Arformoterol 50 mcg QD and placebo MDI
  Interventions: Drug: arformoterol tartrate inhalation solution
- 2 (Experimental): Arformoterol 25 mcg BID and Placebo MDI
  Interventions: Drug: arformoterol tartrate inhalation solution
- 3 (Experimental): Arformoterol 15 mcg BID and placebo MDI
  Interventions: Drug: arformoterol tartrate inhalation solution
- 4 (Active Comparator): Salmeterol MDI 42 mcg BID and placebo inhalation solution
  Interventions: Drug: Salmeterol
- 5 (Placebo Comparator): Placebo MDI and placebo inhalation solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: arformoterol tartrate inhalation solution — arformoterol 50 mcg QD
  Other Names: (R,R)-formoterol
  Arms: 1
Drug: arformoterol tartrate inhalation solution — arformoterol 25 mcg BID
  Other Names: (R,R)-formoterol
  Arms: 2
Drug: arformoterol tartrate inhalation solution — arformoterol 15 mcg BID
  Other Names: (R,R)-formoterol; Brovana
  Arms: 3
Drug: Salmeterol — Salmeterol MDI 42 mcg BID
  Other Names: Serevent MDI
  Arms: 4
Drug: Placebo — Placebo BID
  Arms: 5

SUMMARY:
The purpose of this study is to assess the bronchodilator effect and safety of multiple daily doses of arformoterol administered for 12 weeks as maintenance treatment in patients with COPD

DETAILED DESCRIPTION:
This was a double-blind, double-dummy, randomized, placebo- and active-controlled, multicenter, parallel-group study of adult subjects with COPD. The study was double blinded through the use of both unit dose vial (UDV) and metered-dose inhaler (MDI) placebos, as appropriate. The primary efficacy analysis utilized the placebo control. Secondary analyses of the primary efficacy endpoint utilized the active control, and included comparisons between the placebo and active control. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Be willing to comply with study procedures and visit schedule
* Are at least 35 years of age
* Female subjects >65 years of age must have a serum pregnancy test conducted at Visit 1 and confirmed negative prior to randomization
* Subjects of childbearing potential must be using an acceptable method of birth control. Female subjects who are considered not of childbearing potential must be: documented surgically sterile, OR postmenopausal.
* Have a primary diagnosis of COPD. Diagnosis can be made during the screening process.
* Have a minimum smoking history of 15 pack-years (pack-years = the number of cigarette packs per day times the number of years).
* Have a chest x-ray that is consistent with the diagnosis of COPD and taken <3 months prior to study start
* Able to complete all study questionnaires and logs reliably

Exclusion Criteria:

* Female subject who is pregnant or lactating
* Have participated in an investigational drug study within 30 days prior to study start, or who is currently participating in another investigational drug study
* Subject whose schedule or travel prevents the completion of all required visits
* Are scheduled for in-patient hospitalization, including elective surgery during the trial
* Have life-threatening/unstable respiratory status, including upper or lower respiratory tract infection, within the previous 30 days
* History of asthma or any chronic respiratory disease other than COPD (chronic bronchitis and/or emphysema)
* Have clinically significant cardiac, hepatic, renal, gastrointestinal, endocrine, metabolic, neurologic, or psychiatric disorder that may interfere with successful completion of this protocol
* Have a history of cancer except non-melanomatous skin cancer
* Have a history of lung resection of more than one full lobe
* Requires continuous supplemental oxygen therapy.
* Has had a change in dose or type of any medications for COPD within 14 days prior to the screening visit
* Have a known sensitivity to arformoterol, ipratropium, salmeterol or albuterol or any of the excipients contained in any of these formulations
* Have a history of substance abuse or drug abuse within 12 months, or with a positive urine drug screen
* Are using any prescription drug for which concomitant beta-agonist administration is contraindicated (e.g., beta-blockers)

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 741 (Actual)
Dates: Start 2002-04; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
percent change in trough FEV1 from study baseline to the end of the dosing interval (12 hours post-second dose for the BID treatment arms and 24 hours postdose for the QD treatment arm) over the double-blind period. | Weeks -2, 0, 3, 6, 9, 12

SECONDARY OUTCOMES:
time-normalized area under the percent change from visit predose curve for FEV1 over 12 hours (nAUC0-12-P) | Weeks -2, 0, 3, 6, 9, 12
Peak percent of predicted FEV1 | Weeks -2, 0, 3, 6, 9, 12
time-normalized area under the percent change in FEV1 from study baseline over 12 hours (nAUC0-12-B) | Weeks -2, 0, 3, 6, 9, 12
time-normalized area under the percent change from visit predose curve for FEV1 over 24 hours (nAUC0-24-P) | Weeks -2, 0, 3, 6, 9, 12
time-normalized area under the percent change in FEV1 from study baseline curve over 24 hours (nAUC0-24-B) | Weeks -2, 0, 3, 6, 9, 12
peak percent change in FEV1 from visit predose and study baseline | Weeks -2, 0, 3, 6, 9, 12
time point changes in FEV1; time to onset of response | Weeks -2, 0, 3, 6, 9, 12
time to peak change in FEV1 | Weeks -2, 0, 3, 6, 9, 12
at-home and in-clinic peak expiratory flow rate (PEFR) | Weeks -2, 0, 3, 6, 9, 12
relationship between the plasma concentration values and selected pharmacodynamic parameters | Weeks -2, 0, 3, 6, 9, 12, 13
Supplemental ipratropium bromide MDI and racemic albuterol MDI use | Weeks 0-13
COPD exacerbations and COPD symptom ratings | Weeks 0-13
St. George's Hospital Respiratory Questionnaire | Weeks 0, 6, 13
Investigator and Subject Global Evaluations | Weeks -2, 12, 13
Baseline and Transitional Dyspnea Index | Weeks -2, 6, 12
distance walked in six minutes | Weeks -2, 3, 9

CONTACTS AND LOCATIONS:
Locations (64):
- United States (64):
  - Pulmonary & Sleep Associates of Jasper, PC, Jasper, Alabama
  - Pulmonary Associates, PA, Phoenix, Arizona
  - Arizona Clinical Research Center, Inc., Tucson, Arizona
  - Northern California Research Corp., Fair Oaks, California
  - SARC Research Center, Fresno, California
  - California Research Medical Group, Inc., Fullerton, California
  - Radiant Research-Irvine, Irvine, California
  - West Coast Clinical Trials, Newport Beach, California
  - Center for Clinical Trials, LLC, Paramount, California
  - Advances in Medicine, Rancho Mirage, California
  - Institute of Healthcare Assessment, Inc., San Diego, California
  - San Jose Clinical Research, San Jose, California
  - Allergy & Asthma Medical Group of Diablo Valley, Inc., Walnut Creek, California
  - Colorado Pulmonary Associates, Denver, Colorado
  - Northern Colorado Pulmonary Consultants, PC, Fort Collins, Colorado
  - Physicians Research Center, Inc., Hartford, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - University Clinical Research, DeLand, DeLand, Florida
  - Mt. Sinai Medical Center, Miami Beach, Florida
  - Clinical Pharmacology Services, Tampa, Florida
  - Protocare Trial, Inc., Austell, Georgia
  - Marietta Pulmonary Medicine, Marietta, Georgia
  - Office of Bradley Sakran, MD, PC, O'Fallon, Illinois
  - South Bend Clinic, South Bend, Indiana
  - Family Allergy & Asthma Research Institute, Louisville, Kentucky
  - Cumberland Lung and Sleep Specialists, Somerset, Kentucky
  - Bendel Medical Associates/Research, Lafayette, Louisiana
  - Best Clinical Trials, LLC, New Orleans, Louisiana
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - North Shore Research Associates, Slidell, Louisiana
  - Sunset Medical Research, Sunset, Louisiana
  - University of Maryland-Airways Research Center, Baltimore, Maryland
  - Institute of Asthma and Allergy, Wheaton, Maryland
  - Pro-Medica Clinical Research Center, Boston, Massachusetts
  - ClinSite, Inc., Ann Arbor, Michigan
  - Midwest Chest Consultants, PC, Saint Charles, Missouri
  - MedEx HealthCare Research, Inc., St Louis, Missouri
  - C.A.R.E Clinical Research, St Louis, Missouri
  - Office of Keith Popovich, MD, Butte, Montana
  - Montana Medical Research, LLC, Missoula, Montana
  - VA Medical Center, Omaha, Nebraska
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Pulmonary Medicine, Chapel Hill, North Carolina
  - Charlotte Lung and Health Center, Charlotte, North Carolina
  - Carolina Pharmaceutical Research, Inc., Statesville, North Carolina
  - New Hanover Medical Research, Wilmington, North Carolina
  - New Horizons Clinical Research, Inc., Cincinnati, Ohio
  - COR Clinical Research LLC, Oklahoma City, Oklahoma
  - Allergy Associates Research Center, Portland, Oregon
  - Northeast Clinical Research Centers, Inc., Allentown, Pennsylvania
  - Keystone Clinical Solutions, Altoona, Pennsylvania
  - Philadelphia Health Associates - Adult Medicine, Philadelphia, Pennsylvania
  - Consortium Clinical Research, Ltd., Ridley Park, Pennsylvania
  - Safe Harbor Clinical Research, East Providence, Rhode Island
  - Spartanburg Pharmaceutical Research, Spartanburg, South Carolina
  - Volunteer Research Group, Knoxville, Tennessee
  - Breath of Life Research Institute, Houston, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Pulmonary Associates of Fredericksburg, Inc., Fredericksburg, Virginia
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia
  - Bellingham Asthma, Allergy & Immunology Clinic, Bellingham, Washington
  - University of Wisconsin-Medical School, Madison, Wisconsin